CLINICAL TRIAL: NCT04720651
Title: Prevalence of Calf Muscle Tightness in Asymptomatic Flat Foot Subjects
Brief Title: Calf Muscle Tightness in Flat Foot Subjects
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Hassan Kamel, Teaching Assisstant, Cairo University
Other Study IDs: Calf muscle in flat foot
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Flat Feet
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the current work is to determine the prevalence of calf muscle tightness in asymptomatic flat foot subjects.

DETAILED DESCRIPTION:
Pes planus (Flat foot) deformity is a common chronic foot and ankle condition characterized by flattening of the medial longitudinal arch (MLA), rearfoot valgus and abduction of the midfoot on the hind foot.

A flexible pes planus is caused by tibialis posterior dysfunction, ligament loosening, Achilles tendon shortening, and weakness of the intrinsic foot muscles. These deformations cause plantar flexion and adduction of the talus bone and valgus of the calcaneus bone.

Up to our knowledge:

1. No previous studies investigated whether all flat foot is usually associated with gastrocnemius and soleus muscle tightness or it is a random association.
2. And whether tightness of gastrocnemius and soleus is highly found in all cases of flat foot.

Consequently this study is conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects should have flexible flat foot.
2. Age between 20 and 40 years.
3. Navicular drop of more than 10 mm.
4. Body Mass Index from 18.5 kg/m2 to 29.9 kg/m2.
5. Subjects will sign the written consent form after the aim and methods of the study are explained clearly.

Exclusion Criteria:

1. Subjects with history of foot and ankle surgery, trauma, fracture or dislocation.
2. Subjects with congenital deformities in the ankle and foot.
3. Subjects with systemic or neurologic diseases that could affect lower extremity biomechanics.

Ages: 20 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Subjects with flexible flat foot aged between 20 and 40 years old . They should have navicular drop more than 10 mm and their body mass index is between 18.5 kg/m2 to 29.9 kg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
tightness of the calf muscle | 3 months
  measuring of ankle dorsi flexion range of motion with knee extension and with knee flexion in flat foot subjects with navicular drop more than 1 cm

REFERENCES:
- [Background] Meehan RE, Brage M. Adult acquired flat foot deformity: clinical and radiographic examination. Foot Ankle Clin. 2003 Sep;8(3):431-52. doi: 10.1016/s1083-7515(03)00019-6. PMID 14560897
- [Background] Tome J, Nawoczenski DA, Flemister A, Houck J. Comparison of foot kinematics between subjects with posterior tibialis tendon dysfunction and healthy controls. J Orthop Sports Phys Ther. 2006 Sep;36(9):635-44. doi: 10.2519/jospt.2006.2293. PMID 17017268
- [Background] Van Boerum DH, Sangeorzan BJ. Biomechanics and pathophysiology of flat foot. Foot Ankle Clin. 2003 Sep;8(3):419-30. doi: 10.1016/s1083-7515(03)00084-6. PMID 14560896